CLINICAL TRIAL: NCT06780553
Title: Proteomic Profiling as a Diagnostic Test for Extrahepatic Cholangiocarcinoma on Cytological Samples : Validation of a Proof-of-concept.
Brief Title: Validation of the Proteomic Profiling as a Diagnostic Test for Extra-hepatic Cholangiocarcinoma
Acronym: PROFI-CHOL
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: University of Bordeaux (Other); Plateforme Oncoprot (TBMCore 3427 - US005, Bordeaux Biologie Santé) (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2024/32
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Cholangiocarcinoma
Keywords: cholangiocarcinoma; biopsy; diagnosis; proteomic profiling; proteomic
MeSH Terms: conditions — Cholangiocarcinoma; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected cholangiocarcinoma: Patient with biliary stenosis of undetermined origin who has had an endo-biliary cytological sample (biopsy and/or brushing) for suspected cholangiocarcinoma
  Interventions: Diagnostic Test: Proteomic profiling

INTERVENTIONS:
Diagnostic Test: Proteomic profiling — Proteomic profiling as a diagnostic tool in the face of suspected extrahepatic cholangiocarcinoma stenosis

SUMMARY:
The study aims to valide a proof of a concept of the proteomic profiling as a diagnostic tool for bile duct stenosis suspicious of cholangiocarcinoma. The main objective is to evaluate the addition of proteomic profiling to the conventional histological diagnosis of endo-biliary cytological sampling of biliary stenosis, compared with cytological sampling alone. With the addition of proteomic profiling to the conventional histological diagnostic technique, an overall diagnostic sensitivity of 80% is expected

DETAILED DESCRIPTION:
Cholangiocarcinoma is a cancer with an increasing incidence and a poor prognosis (< 5% of all stages at 5 years). The extra-hepatic form is the most common and is rarely resectable at diagnosis (30% of cases). This is due to the late onset of symptoms, which often indicate that the disease is too advanced. It can also be explained by the diagnostic difficulties encountered with this cancer. In fact, the reference diagnostic technique is histological testing on endo-biliary cytological samples taken by biopsy and/or brushing during catheterisation of the bile ducts or by interventional radiology. The problem is that the sensitivity of this test is of the order of 50%, with an additional diagnostic uncertainty of the order of 20 to 30%, due to cellular atypia that are not sufficiently clear to confirm a cancerous pathology, although it is not possible to exclude it. This leads to diagnostic error and delay, repeated invasive examinations and sometimes major surgery for stenoses that are ultimately benign when the surgical decision has been taken without a reliable histological result. Additional diagnostic techniques are needed to diagnose a suspected extrahepatic cholangiocarcinoma stenosis, particularly at the molecular level using proteomics and, above all, proteomic profiling. Proteomic profiling enables a patient's diagnosis to be oriented towards a profile (benign or malignant) by comparing the proteins identified in formalin-fixed, paraffin-embedded tissue (cytological sample) with a set of proteins identified within a reference diagnostic signature obtained from previously analysed benign and malignant samples. Within Inserm Unit 1312 - Team 3, a proof of concept for proteomic profiling has been developed as a diagnostic tool in the face of suspected extrahepatic cholangiocarcinoma stenosis, with the development of a diagnostic signature. The aim of this project is to validate this proof of concept on a large retrospective monocentric cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient with biliary stenosis of undetermined origin who has had an endo-biliary cytological sample (biopsy and/or brushing) for suspected cholangiocarcinoma, fixed in formalin and included in paraffin with at least 1 year of follow-up.
* No objection to re-use of data

Exclusion Criteria:

* Absence of cellular material usable in proteomics on residual histological block
* Presence of pancreatic adenocarcinoma demonstrated on cytological sampling, definitive histology after surgical resection and/or clinical-morphological follow-up of at least one year.
* Patient under legal protection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with biliary stenosis of undetermined origin who has had an endo-biliary cytological sample (biopsy and/or brushing) for suspected cholangiocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the proteomic profiling | Baseline
  Sensitivity of the proteomic profiling test combined with conventional histological diagnosis, compared with the sensitivity of the conventional histological diagnostic test alone.

SECONDARY OUTCOMES:
Accuracy of the proteomic profiling | Baseline
  The accuracy of the proteomic profiling associated with the conventional histological test (specificity, positive predictive value, negative predictive value)
Molecular pathway of cholangiocarcinogenesis | Baseline
  Identification of the molecular pathway of cholangiocarcinogenesis using Gene Set Enrichment Analysis

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Pessac, France

IPD SHARING:
Plan to Share IPD: No